CLINICAL TRIAL: NCT01871363
Title: Phase II Study of Preoperative IMRT Combined With Capecitabine and Bevacizumab in Locally Advanced Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hua Ren, Attending Radiation oncologist, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-027
Record Dates: First submitted 2013-05-19; First posted 2013-06-06 (Estimated); Last update posted 2013-06-06 (Estimated); Status verified 2013-06

CONDITIONS: Locally Advanced Malignant Neoplasm
Keywords: Preoperative Chemoradiotherapy; Bevacizumab; Locally Advanced Rectal Cancer
MeSH Terms: interventions — Chemoradiotherapy; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- preoperative chemoradiation (Experimental): * radiotherapy: 50 Gy to the pelvis (25x 2 Gy on days 1-35, excluding weekends) .IMRT planing and technique with high energy photons will be used. All fields will be treated daily. Multileaf collimators will be used to shape individual radiation fields. Patients will be irradiated in a prone position with a full bladder and by using belly board to minimize exposure of the small bowel.
  * capecitabine 825 mg/m² p.o. twice daily on days 1-35 (including weekends),
  * bevacizumab: at dose 5 mg/kg on days -1, 15,31.
  * Radical surgery (TME): to be undertaken ideally 6-8 weeks following completion of chemoradiation.
  Interventions: Radiation: chemoradiation

INTERVENTIONS:
Radiation: chemoradiation — * radiotherapy: 50 Gy to the pelvis (25x 2 Gy on days 1-35, excluding weekends) .IMRT planing and technique with high energy photons will be used. All fields will be treated daily. Multileaf collimators will be used to shape individual radiation fields. Patients will be irradiated in a prone position with a full bladder and by using belly board to minimize exposure of the small bowel.
  * capecitabine 825 mg/m² p.o. twice daily on days 1-35 (including weekends),
  * bevacizumab: at dose 5 mg/kg on days -1, 15, 31.
  * Radical surgery (TME): to be undertaken ideally 6-8 weeks following completion of chemoradiation.
  Other Names: Preoperative Radiotherapy With Capecitabine and Bevacizumab

SUMMARY:
Pathological complete response, (pCR) correlates with a favourable overall prognosis in locally advanced rectal cancer patients underwent preoperative chemoradiation, so obtaining a pCR might be beneficial. The aim of the study is to investigate safety and efficacy of preoperative IMRT combined with bevacizumab and capecitabine. primary endpoint is pathological complete remission rate.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with histologically proven adenocarcinoma of the rectum ,T3/4 or any node positive disease (clinical stage according the TNM classification system)
* No evidence of metastatic disease.
* Age 18 - 65 years
* Kps 80-100
* No prior radiotherapy, chemotherapy or any targeting therapy for rectal cancer
* Normal hematological, hepatic and renal function, Ability to swallow tablets
* Signed informed consent
* Patients must be willing and able to comply with the protocol for duration of the study

Exclusion Criteria:

* Malignancy of the rectum other than adenocarcinoma

  * Other co-existing malignancy or malignancy within the past 5 years, with the exception of adequately treated in situ carcinoma of the cervix or basal cell carcinoma of the skin
  * Significant heart disease (uncontrolled hypertension despite of medication (> 150/100 mmHg), NYHA class III or IV heart disease,unstable angina or myocardial infarction within the past 1 year prior the study entry, history of significant ventricular arrhythmia requiring treatment)
  * Evidence of active peptic ulcer or upper GI bleeding
  * Evidence of bleeding diathesis or coagulopathy
  * Patients receiving a concomitant treatment with drugs interacting with capecitabine such as flucitosine, phenytoin, or warfarin
  * Known hypersensitivity to biological drugs
  * Treatment with any investigational drug within 30 days before beginning treatment with the study drug
  * Pregnant or lactating patient

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission rate (pCR) | after pathological examination of surgical speciments (6-8 weeks after chemoradiation)
  A TME surgery will be done 6-8 weeks after concurrent chemoradiation, pathological examination of surgical speciments will be show Pathological complete remission rate (pCR)

SECONDARY OUTCOMES:
Acute and late toxicity | Toxicity/safety:during preoperative treatment, early and late postoperative follow up
  Acute toxicities will be assessed every week during chemoradiation period , one week before surgery(6 weeks after chemoradiation) and every 3 months after surgery for 2 years.
  late toxicites will be assessed every 6 months from the third year after surgery.

OTHER OUTCOMES:
Disease-free survival | 3 year afte concurrent chemoradiation
  Followup will be done every 3 months in first 2 years, and every 6 months after 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jin, proffessor, Study Chair — Dept of Radiation oncology, Cancer hospital, CAMS
Locations (1):
- Cancer Hospital, CAMS, Beijing, China